CLINICAL TRIAL: NCT02433002
Title: Accuracy of Glomerular Filtration Rate Estimation Using Creatinine & Cystatin C & Albuminuria for Monitoring Disease Progression in Patients With Stage 3 Chronic Kidney Disease: Prospective Longitudinal Study in a Multi-ethnic Population
Brief Title: Accuracy of Glomerular Filtration Rate (GFR) Estimation Using Creatinine and Cystatin C and Albuminuria
Acronym: eGFR-C
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University of Birmingham (Other)
Collaborators: East Kent Hospitals University NHS Foundation Trust (Other Government); National Institute for Health Research, United Kingdom (Other Government)
Responsible Party: Sponsor
Other Study IDs: RG_13-176; ISRCTN42955626 (Registry Identifier: ISRCTN); 11/103/01 (Other Grant/Funding Number: NIHR HTA); 15268 (Other: UKCRN); 13/LO/1349 (Other: NRES Committee: South East Coast - Surrey)
Record Dates: First submitted 2015-04-15; First posted 2015-05-04 (Estimated); Last update posted 2021-09-29 (Actual); Status verified 2021-09

CONDITIONS: Chronic Kidney Diseases
Keywords: eGFR; CKD; Cystatin; Creatinine; Albuminuria
MeSH Terms: conditions — Renal Insufficiency, Chronic; Albuminuria

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum/plasma and urine will be stored for potential analysis of future markers.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Main study: 1300 participants will undergo baseline (month 0) and final (month 36) reference GFR, estimated GFR (eGFR) and urinary albumin-to-creatinine ratio (ACR) tests. Additionally they will provide ACR and eGFR tests at 6-monthly intervals.
- Sub-study of patterns of progression: A subset of the cohort (n=375) will receive annual reference GFR tests.
- Biological variability study: In a further sub-study 20 participants will undergo the reference test four times over four weeks.

SUMMARY:
The eGFR-C study will assess the accuracy of current and alternative tests of kidney function against a reference test in people with moderate (stage 3) chronic kidney disease (CKD).

DETAILED DESCRIPTION:
The eGFR-C study will assess the accuracy of current and alternative tests of kidney function against a reference test in people with moderate (stage 3) CKD. Participants will be recruited from hospital clinics and General Practitioner (GP) practices at six major United Kingdom (UK) centres.

The best measure of kidney function is accepted to be the glomerular filtration rate (GFR), which measures the ability of the kidney to filter blood and is widely used in clinical practice. A low GFR suggests poor kidney function. An estimate of GFR can be obtained from a simple blood test.

Participants will undergo reference GFR testing at study entry with a second follow-up reference test three years later. The reference test involves injecting a small amount of iohexol into a vein and taking blood samples over the next 4 hours to see how quickly the iohexol disappears from the blood stream as a result of glomerular filtration. The rate at which iohexol disappears is equivalent to the level of kidney function. Blood tests for monitoring kidney function, including testing for creatinine and cystatin C, and measurement of urinary albumin will be done every six months during the study period.

Iohexol measured GFR will be accepted as the reference ('gold standard') measure of kidney function against which each GFR-estimating equations will be compared. The alternative estimated measures of GFR, derived from measuring substances (creatinine and cystatin C) in the blood, will be compared against the reference test. An important outcome is how much the reference test changes over the three years of the study, and how well the surrogate measures reflect this change.

The investigators will also collect accurate test cost data for subsequent cost-effectiveness analysis (e.g. do the relative costs of the tests justify any change in practice due to improved performance of one test compared to another?).

ELIGIBILITY:
Inclusion Criteria:

* Patients with stage 3 CKD (GFR 30-59 mL/min/1.73 m2) as defined internationally, diagnosed using MDRD/CKDEPI eGFR (at least two consecutive test results in this range at least 90 days apart, with the most recent test in the last 12 months)
* Aged 18 years or over
* Written informed consent

Exclusion Criteria:

* History of untoward reactions to iodinated contrast media or allergy to topical iodine
* Episode of acute kidney injury in previous 6 months (as defined by the Acute Kidney Injury Network criteria)
* Amputation of whole or part-limb
* Pregnant or breastfeeding
* Known current alcohol or drug abuse
* Kidney transplant recipient
* Any condition with an expected survival of less than study duration
* Inability to comply with study schedule and follow-up
* Inability to provide informed consent e.g. due to cognitive impairment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults with stage 3 CKD.
Sampling Method: Non-Probability Sample
Enrollment: 1249 (Actual)
Dates: Start 2014-04-08 (Actual); Primary Completion 2020-01-31 (Actual); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Percentage of estimated Glomerular Filtration Rate values within 30% of 'true' Glomerular Filtration Rate | Baseline
  The accuracy of Glomerular Filtration Rate (GFR) estimating equations is commonly expressed as the P30 value, the percentage of estimated GFR values within 30% of 'true' GFR.
  The eGFR-C study will estimate and compare the accuracy and precision of GFR-estimating equations based on the Modification of Diet in Renal Disease (MDRD) equation and three Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) equations using either creatinine or cystatin C or a combination of both in people with stage 3 Chronic Kidney Disease (CKD), expressed as the P30 value.

CONTACTS AND LOCATIONS:
Overall Officials: Edmund Lamb, PhD, FRCPath, Principal Investigator — East Kent Hospitals University NHS Foundation Trust
Locations (6):
- United Kingdom (6):
  - Derby Hospitals NHS Foundation Trust (Royal Derby Hospital), Derby, Derbyshire
  - King's College Hospital NHS Foundation Trust, London, Greater London
  - Salford Royal NHS Foundation Trust (Salford Royal Hospital), Salford, Greater Manchester
  - East Kent Hospitals NHS Trust (Kent & Canterbury Hospital), Canterbury, Kent
  - University Hospitals of Leicester NHS Trust (Leicester General Hospital), Leicester, Leicestershire
  - University Hospital Birmingham NHS Trust (Queen Elizabeth Hospital Birmingham), Birmingham, West Midlands

REFERENCES:
- [Background] Lamb EJ, Brettell EA, Cockwell P, Dalton N, Deeks JJ, Harris K, Higgins T, Kalra PA, Khunti K, Loud F, Ottridge RS, Sharpe CC, Sitch AJ, Stevens PE, Sutton AJ, Taal MW; eGFR-C study group. The eGFR-C study: accuracy of glomerular filtration rate (GFR) estimation using creatinine and cystatin C and albuminuria for monitoring disease progression in patients with stage 3 chronic kidney disease--prospective longitudinal study in a multiethnic population. BMC Nephrol. 2014 Jan 14;15:13. doi: 10.1186/1471-2369-15-13. PMID 24423077
- [Derived] Rowe C, Sitch AJ, Barratt J, Brettell EA, Cockwell P, Dalton RN, Deeks JJ, Eaglestone G, Pellatt-Higgins T, Kalra PA, Khunti K, Loud FC, Morris FS, Ottridge RS, Stevens PE, Sharpe CC, Sutton AJ, Taal MW, Lamb EJ; eGFR-C Study Group. Biological variation of measured and estimated glomerular filtration rate in patients with chronic kidney disease. Kidney Int. 2019 Aug;96(2):429-435. doi: 10.1016/j.kint.2019.02.021. Epub 2019 Mar 7. PMID 31084924
- See also: Plain English summary — https://www.birmingham.ac.uk/research/bctu/trials/renal/egfr-c/participants/index.aspx
- See also: Study website — http://www.birmingham.ac.uk/egfr-c